CLINICAL TRIAL: NCT04524208
Title: CABONEN - A Phase II Trial of Cabozantinib in Patients With Advanced, Low Proliferative NEN G3
Brief Title: A Trial of Cabozantinib in Patients With Advanced, Low Proliferative NEN G3
Acronym: CABONEN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karsten Gavenis (Other)
Responsible Party: Sponsor-Investigator, Karsten Gavenis, Project Manager, University Medical Center Goettingen
Organization: University Medical Center Goettingen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02679
Record Dates: First submitted 2020-08-18; First posted 2020-08-24 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Carcinoma
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment-Arm (Experimental)
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib is administered orally at the dose of 60 mg per day..

SUMMARY:
The main objective of this clinical trial represents the evaluation of efficacy of the tyrosine kinase inhibitor Cabozantinib in patients with NEN G3 with a proliferation rate of Ki67 20 - 60%.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically confirmed diagnosis of neuroendocrine neoplasia;
2. Tumor proliferation rate has to be between Ki67 20% to 60% (local assessment);
3. Male, female, or diverse patients aged > 18 years without upper age limit;
4. At least one measurable tumor lesions in CT or MRI scan;
5. Newly diagnosed or progressive disease assessed per RECIST criteria 1.1;
6. Patients must have a performance status of ECOG 0-2;
7. Patients must have a life expectancy of more than 3 months;
8. Hb> 9 mg/dl;
9. platelets >80T/µl;
10. white blood cells >3T/μL;
11. total bilirubin <3mg/dl;
12. AST and ALT <4xN;
13. Serum creatinine <2mg/dl, eGFR >40mL/min/1.73m2;
14. BUN <5xN;
15. lipase <3xN;
16. albumin ≥2.8 g/dL;
17. PT/PTT ≤ 1.5 × ULN;
18. urine protein: creatinine ratio ≤ 1;
19. Written informed consent obtained according to international guidelines and local laws;
20. Ability to understand the nature of the trial and the trial related procedures and to comply with them;

Exclusion Criteria:

1. Patients younger than 18 years;
2. Patients with Mixed Neuroendocrine-Non-neuroendocrine Neoplasia (MINEN);
3. Patients with former treatment with TKI or VEGF receptor antagonist;
4. Patients with additional malignancy <5 years in medical history (exclusion: non-invasive skin cancer);
5. Patients with symptomatic brain metastases;
6. Patients with Known HIV infection, infectious hepatitis (type A, B or C) or another uncontrolled infection;
7. Patients with Known hypersensitivity to Cabozantinib or contraindications for treatment with Cabozantinib according to Summary of Product Characteristics (SmPC);
8. Patients with class III or IV congestive heart failure;
9. Patients with QTc more than 500 ms or 140% of normal range according to age;
10. Patients with uncontrolled hypertension;
11. Patients with severely impaired lung function;
12. Patients with history of organ transplant (exclusion: cornea transplantation);
13. Patients with clinical apparent acute or chronic gastric ulceration;
14. Patients with history of hemophilia;
15. Patients with surgery at the GI tract within the last 12 weeks;
16. Patients with patients with uncontrolled inflammatory bowel disease;
17. Simultaneous participation in other interventional trials which could interfere with this trial; simultaneous participation in registry and diagnostic trials is allowed
18. Patient without legal capacity who is unable to understand the nature, significance and consequences of the trial;
19. Previous participation in this trial
20. concomitant use of therapeutic anticoagulation or strong CYP3A4 inducers or inhibitors (e.g. amiodarone);
21. Known or persistent abuse of medication, drugs or alcohol;
22. Person who is in a relationship of dependence/employment with the sponsor or the investigator;
23. Patients who cannot give informed consent;
24. Current or planned pregnancy, nursing period;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of Cabozantinib treatment via DCR after 6 months. | 6 months
  Disease control rate (DCR) 6 months after treatment start .

SECONDARY OUTCOMES:
Evaluate short- and long term efficacy of Cabozantinib treatment via DCR. | 12 months
  DCR 3 and 12 months after treatment start.
Evaluate short- and long term efficacy of Cabozantinib treatment via ORR. | 12 months
  Objective response rate (ORR) 3, 6 and 12 months after treatment start and best objective response rate.
Evaluate short- and long term efficacy of Cabozantinib treatment via PFS. | 24 months
  Progression free survival (PFS).
Evaluate short- and long term efficacy of Cabozantinib treatment via OS. | 24 months
  Overall survival (OS).
Evaluate exposure time. | 12 months
  Time on drug (TOD).
Assess quality-of-life during and after Cabozantinib treatment. | 15 months
  EORTC QLQ-C30 Quality of Life Questionnaire monthly for 12 months after treatment start and after 15 months. Different questions regarding Quality of Life on a scale of 1 - 4. The lower the numbers, the better the quality of Life.

OTHER OUTCOMES:
Safety of Cabozantinib via AE and SAE assessment. | 24 months
  Adverse events and serious adverse events will be assessed in contingency tables.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander König, PD Dr., Principal Investigator — University Medical Center Göttingen
Locations (15):
- Medizinische Universität Wien, Vienna, Austria
- Germany (14):
  - University Medical Center Göttingen, Göttingen, Lower Saxony
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Halle, Halle
  - Asklepios St. Georg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Heidelberg, Heidelberg
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Johannes-Wesling-Klinikum Minden, Minden
  - Klinikum Ulm, Ulm
  - Universitätsklinik Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No